CLINICAL TRIAL: NCT03974490
Title: Effect of Rhythmic Auditory Stimulation on Balance and Gait Parameters in Stroke Patients
Brief Title: Effect of RAS on Balance and Gait After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Sociosanitari Mutuam Girona (Other)
Responsible Party: Principal Investigator, Samira Gonzalez Hoelling, Principal Investigator, Physiotherapist, Hospital Sociosanitari Mutuam Girona
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mutuam_Girona_04_19
Record Dates: First submitted 2019-04-11; First posted 2019-06-05 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Stroke; Gait, Hemiplegic; Gait Disorders, Neurologic
Keywords: rhythm; musicotherapy; balance; gait; stroke; physiotherapy
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): 2 hours from Monday to Saturday, conventional physiotherapy: strengthening, stretching, dual task training.
  3 Times a week, intervention: Start with global body warming, 15 minutes, following the rhythm marked by the metronome. Central part of the session, 60 minutes, with rhythmic auditory stimulation exercises and music. Closure of the session, 15 minutes, round of impressions.
  Interventions: Other: Rhythmic auditory stimulation
- Historical control group (No Intervention): 2 hours from Monday to Saturday, conventional physiotherapy: strengthening, stretching, dual task training.

INTERVENTIONS:
Other: Rhythmic auditory stimulation — Rhythmic auditory stimulation 3 times in a week, and 2 hours of physiotherapy 6 days in a week.
  Arms: Intervention Group

SUMMARY:
A rhythmic auditory stimulation intervention may be beneficial in order to improve movement parameters after stroke. Reviews argue that more randomized controlled trials with a control group are needed. Main objective: Evaluate the effect of a rhythmic auditory stimulation on the quality of balance and gait parameters in people with stroke. Methodology: quasi-experimental study. The study has been approved by the hospital ethics committee.

DETAILED DESCRIPTION:
A rhythmic auditory stimulation (RAS) intervention may be beneficial in order to improve the parameters of the post-stroke movement: increase of the speed of the walk, improvement in the width of the step with the affected side, improvement of the walking index dynamics (Dynamic Gait Index), improvement in cadence and improvement in the static balance.

Current systematic reviews argue that more randomized controlled trials with a control group are needed.

Main objective: To evaluate the effect of a rhythmic auditory stimulation on the quality of progress and balance in people with stroke.

Methodology: experimental group will be done between 2019 and 2020 and historical control group of the years 2017 and 2018. Experimental group will do 3 sessions in a week of RAS, and daily 2 hours of physiotherapy except of Sundays. Control group received 2 hours daily of physiotherapy, except Sundays.

The study has been approved by the hospital ethics committee.

ELIGIBILITY:
Inclusion Criteria:

* Had a stroke in the last 3 weeks
* Rankin 3-4
* Barthel before stroke: >85
* Tinetti < 23

Exclusion Criteria:

* Patient can walk independently (Functional Ambulation Category >3)
* Global and/or mixed aphasia
* Glasgow < 10
* Mini-Mental State Examination < 24
* Posterior cerebral artery stroke
* Gait and/or balance disorders before stroke (parkinsons disease, neurodegenerative diseases)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Balance | At baseline, 20 days after baseline and 40 days after baseline
  Change in balance using the Mini Best Test
Balance | At baseline, 20 days and 40 days after baseline
  Change in balance using the Tinetti Test
Gait | At baseline, 20 days after baseline and 40 days after baseline
  Change in gait using the Tinetti Test
Gait | At baseline, 20 days and 40 days after baseline
  Change in gait using the Timed Up&Go Test
Gait parameters | At baseline, 20 days after baseline and 40 days after baseline
  Change in step length using a measure tape
Gait parameters | At baseline, 20 days and 40 days after baseline
  Change in stride length using a measure tape
Gait parameters | At baseline, 20 days after baseline and 40 days after baseline
  Change in cadence using a stopwatch
Gait Functionality | At baseline and 40 days after baseline
  Change in gait functionality using the Functional Ambulatory Category

CONTACTS AND LOCATIONS:
Overall Officials: Samira Gonzalez, Principal Investigator — Hospital Sociosanitari Mutuam Girona
Locations (1):
- Hospital Sociosanitari Mutuam Girona, Girona, Spain

REFERENCES:
- [Derived] Gonzalez-Hoelling S, Bertran-Noguer C, Reig-Garcia G, Suner-Soler R. Effects of a Music-Based Rhythmic Auditory Stimulation on Gait and Balance in Subacute Stroke. Int J Environ Res Public Health. 2021 Feb 19;18(4):2032. doi: 10.3390/ijerph18042032. PMID 33669715